CLINICAL TRIAL: NCT07239349
Title: Investigating Whether Preoperative Use of Acne Face Wash for Cleansing the Face, Neck, and Chest Helps Reduce the Contamination Rate of Cutibacterium Acnes in Arthroscopic Rotator Cuff Repair Surgery
Brief Title: Acne Face Wash for Reducing the Contamination Rate in Arthroscopic Rotator Cuff Repair Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 202510005RINA
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Rotator Cuff Tears of the Shoulder
Keywords: rotator cuff tear; arthroscopy; benzoyl peroxide; Cutibacterium acnes
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Use soap to wash shoulder before surgery
- Acne face wash (Experimental): Use acne face wash to clean shoulder before surgery
  Interventions: Other: Acne face wash

INTERVENTIONS:
Other: Acne face wash — Use acne face wash to clean shoulder before surgery
  Arms: Acne face wash

SUMMARY:
Previous studies have shown that even when following standard sterilization protocols, the positive culture rate of Cutibacterium acnes can still be as high as 30%. In recent years, several studies have reported that preoperative skin preparation of the shoulder, such as applying benzoyl peroxide (BPO) to the skin, can effectively reduce the cutaneous bacterial load of C. acnes and even decrease its incidence in the shoulder joint or surgical sutures after surgery. However, most of the existing studies have focused on arthroplasty, and robust evidence regarding contamination in rotator cuff surgery remains lacking. Therefore, this study aims to investigate whether preoperative skin preparation with a 10% BPO acne cleanser can effectively reduce contamination in rotator cuff surgery. The findings will help guide future clinical practice in preoperative preparation. This study will adopt a prospective randomized design. Patients will be randomly assigned (using a random number table) into two groups: the control group and the BPO cleanser group. All patients will receive instructions on preoperative skin cleansing. Patients in the control group will follow the current routine practice in our institution, cleansing the surgical site (shoulder) with soap or body wash. Patients in the BPO group, in addition to routine preoperative instructions, will receive specific guidance on cleansing the shoulder and surrounding skin. They will be provided with a 10% BPO acne cleanser and instructed to use it on the shoulder and surrounding area during bathing the day before surgery. After surgical disinfection, skin samples will be collected for bacterial culture. In addition, a segment of surgical suture will be obtained postoperatively for bacterial culture.

ELIGIBILITY:
Inclusion Criteria:

* rotator cuff tear
* scheduled for arthroscopic rotator cuff repair surgery

Exclusion Criteria:

* history of shoulder fracture
* previous shoulder surgeries
* tatoo on the shoulder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-11-18 (Estimated); Primary Completion 2026-11-18 (Estimated); Study Completion 2027-11-18 (Estimated)

PRIMARY OUTCOMES:
Suture culture results | Right after the surgery

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No